CLINICAL TRIAL: NCT00039962
Title: Thymosin Plus PEG-Interferon in Hepatitis C Patients With Cirrhosis Who Did Not Respond to Interferon or Interferon Plus Ribavirin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SciClone Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ta1-CHC-2K0804
Record Dates: First submitted 2002-06-17; First posted 2002-06-19 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Hepatitis C; Hepatitis C, Chronic
Keywords: hepatitis C; hepatitis C, chronic; cirrhosis, liver
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Liver Cirrhosis | interventions — Thymalfasin; peginterferon alfa-2a

INTERVENTIONS:
Drug: thymalfasin (thymosin alpha 1)
Drug: PEGinterferon alfa-2a

SUMMARY:
Chronic hepatitis C infection is one of the leading causes of chronic liver disease in the United States. Approximately one-third of patients with hepatitis C infection develop cirrhosis of the liver, which can lead to liver failure or liver cancer. The current treatment for hepatitis C infection in previously untreated patients is successful in only about half of patients. There is no established therapy for non-responders.

This is a randomized, double-blinded, multicenter trial to determine the effectiveness of thymosin alpha 1 (thymalfasin) 1.6 mg twice weekly plus PEGinterferon alfa-2a 180 ug/wk compared to placebo plus PEGinterferon alfa-2a in adults with chronic hepatitis C with early cirrhosis or progression to cirrhosis who are non-responders to previous treatment with interferon or interferon plus ribavirin. The definition of non-response requires a positive HCV RNA test at the end of a course of at least 12 weeks of therapy. Patients will receive treatment for 12 months, and will be followed-up for a further 6 months after the end of therapy

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent.
* Age over 18 years old.
* Presence of HCV RNA measured by qualitative PCR.
* Nonresponder to a previous course of therapy with either IFN alone or IFN plus ribavirin. The patient must have been treated for at least 3 months (12 weeks).
* Washout period of at least 6 months from previous therapy with IFN alone or IFN plus Ribavirin.
* Liver biopsy consistent with cirrhosis or progression to cirrhosis (METAVIR fibrosis score 3 to 4) due to chronic hepatitis C within the last 12 months before treatment starts, and at least 6 months after the end of the prior failed therapy.
* Cirrhosis classified as Child-Pugh "A" (no more than 6 points).
* Compensated liver disease with prothrombin time prolonged less than 3 seconds over control, total bilirubin < 2 mg/dl, and no history of hepatic encephalopathy, bleeding varices or a history of detection of stigmata of recent bleeding on existing varices or ascites.
* Ultrasound, CT scan, or MRI of the liver within 3 months of entry negative for HCC.
* Hematocrit > 30%, platelet count > 75,000, WBC > 2,500, and absolute neutrophil cell count > 1,500.
* Adequate renal function as demonstrated by serum creatinine level < 2.0 mg/dl.
* Normal TSH or adequately controlled thyroid function.
* If the patient is a woman, she is using a definitive method of birth control in consultation with her physician, or is surgically sterile, or post-menopausal.

Exclusion criteria:

* Use of systemic corticosteroids within 6 months of entry.
* Evidence of drug-induced liver injury.
* Current use of any drug known to have or suspected of having therapeutic activity in hepatitis C, or any immunosuppressive drug (including corticosteroids).
* Evidence of any other liver disease including hepatitis B, hepatitis delta, alcoholic liver disease, primary biliary cirrhosis, sclerosing cholangitis, autoimmune hepatitis, hemochromatosis, alpha 1-antitrypsin deficiency, or Wilson's disease.
* Alpha-fetoprotein > 200 ng/mL.
* Child-Pugh "B" or "C" cirrhosis (score of 7 or more points), either currently or at any occasion in the past.
* Decompensated liver disease based on a history of hepatic encephalopathy, bleeding varices or a history of detection of stigmata of recent bleeding on existing varices, or ascites.
* HIV infection diagnosed by HIV seropositivity and confirmed by Western blot.
* Concomitant or prior history of malignancy other than curatively treated skin cancer or surgically cured in situ carcinoma of the cervix.
* Active infectious process other than HCV that is not of a self-limited nature.
* Rheumatoid arthritis or other autoimmune disease (serum ANA > 1:160.).
* Pregnancy as documented by a urine pregnancy test.
* Alcohol or intravenous drug abuse within the previous 1 year.
* Chronic use of methadone.
* Patients who are poor medical risk or who have any non-malignant systemic disease that, in the opinion of the investigator, would make it unlikely that the patient could complete the protocol.
* Patients with a history of severe depression that required either hospitalization or electroshock therapy; or depression associated with suicide attempt.
* Patients with significant pre-existing cardiac or pulmonary disease.
* Recipients of transplants.
* Patients with uncontrolled seizure disorder.
* Any indication that the patient would not comply with the conditions of the study protocol.
* Previous treatment with thymosin alpha 1.
* Patients with known hypersensitivity to IFN a.
* Simultaneous participation in another investigational drug study, or participation in any clinical trial involving investigational drugs within 3 months of study entry.
* Family history of intracerebral hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2002-05

CONTACTS AND LOCATIONS:
Locations (56):
- United States (54):
  - University of Alabama - Knollwood Physician's Group, Mobile, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Gastroenterology Associates of East Bay Medical Group, Berkeley, California
  - Scripps Clinic, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Huntington Memorial Hospital, Pasadena, California
  - Kaiser Permanente, Sacramento, California
  - University of California, Davis Medical Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - San Mateo Medical Center, San Mateo, California
  - Kaiser Permanente, Santa Clara, California
  - Arapahoe Gastroenterology, Littleton, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University Of Miami Center for Liver Diseases, Miami, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Center for Digestive and Liver Health, Savannah, Georgia
  - Idaho Gastroenterology Associates, Meridian, Idaho
  - University of Chicago Hospital & Clinic, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - LSU Healthcare Network, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Endoscopic Microsurgery Associates, Towson, Maryland
  - New England Medical Center, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mississippi Gastrointestinal Associates, Jackson, Mississippi
  - Bradley Freilich MD, LLC, Kansas City, Missouri
  - VAMC, Kansas City, Missouri
  - North Shore University Hospital, Manhasset, New York
  - NYU Gastroenterology & Hepatology, New York, New York
  - VA Harbor HealthCare System, New York, New York
  - Carolinas Center for Liver Disease, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Metro Health Medical Ctr., Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Jefferson University Physicians, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Advanced Clinical Research, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Gastroenterology, Memphis, Tennessee
  - Austin Gastroenterology PA, Austin, Texas
  - Baylor University Medical Ctr., Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Baylor, VAMC, Houston, Texas
  - Metropolitan Research, Fairfax, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Ponce School of Medicine, Ponce
  - Fundacion de Investigacion de Diego, Santurce